CLINICAL TRIAL: NCT02862366
Title: Role of the Circulating Procoagulants Microparticles in the Hypercoagulability of Chronic Philadelphia Negative Myeloproliferative Neoplasms
Brief Title: Role of the Circulating Procoagulants Microparticles in the Hypercoagulability of MNP Ph1-
Acronym: MICROP-SMP
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0004
Record Dates: First submitted 2016-08-02; First posted 2016-08-11 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-08

CONDITIONS: Myeloproliferative Neoplasm
Keywords: myeloproliferative neoplasms; Circulating Procoagulants Microparticles
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Primary Myelofibrosis (PMF): Blood sampling during routine visit
  Interventions: Other: Blood sampling
- Essential thrombocytosis (ET): Blood sampling during routine visit
  Interventions: Other: Blood sampling
- Polycythemia vera (PV): Blood sampling during routine visit
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling every 6 month following the routine calendar of visit

SUMMARY:
Patients with myeloproliferative neoplasms Philadelphia chromosome negative (MPNsPh1-) such as Essential thrombocytosis (ET), Polycythemia vera (PV) and Primary Myelofibrosis (PMF) have a higher risk of arterial or deep-vein thrombosis. This is responsible for a significant increase in mortality (up to 31% of increase in thrombosis risk in ET). Cellular inflation and blood hyperviscosity, resulting from these diseases, fail to account for these thromboses, as more than 50% of thrombotic complications happen under adapted antineoplastic drug treatment.

These last years, cellular microparticles (MPs) have been shown to play a major role in thrombogenesis. MPs are generated by apoptosis or the activation of malignant cells, platelets, endothelial cells or monocytes. They are fragments of plasma membrane, smaller than 1 µm, rich in phosphatidylserine, which can express the tissue factor and serve as support for the coagulation factors. Increase in the plasma concentration of procoagulant platelet microparticles has been demonstrated in other thrombotic diseases (acute coronary syndrome, disseminated intravascular coagulation DIC, etc.). The working hypothesis is that platelet microparticles are involved in the hypercoagulability of MPNs patients.

ELIGIBILITY:
Inclusion Criteria for MNPs patients:

* Age > 18
* Establish MNPs Phi- diagnosis (ET, PV, MFP)
* Consent to participate

Inclusion Criteria for healthy volunteers:

* Healthy volunteers matched in age, sex with the MNPs patients, with a normal complete blood and platelet count
* No personal thromboembolic history
* No known thromboembolic risk factor : thrombophilia, cancers, and other disease associated with a thrombotic risk (Atrial fibrillation, etc.)
* Not pregnant
* Non smoker
* For women, no hormonal contraceptives

Exclusion Criteria for MNPs patients:

* Pregnancy
* Patient unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ET, PV or PMF. Healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2010-10; Primary Completion 2016-01-25 (Actual); Study Completion 2016-01-25 (Actual)

PRIMARY OUTCOMES:
Comparison of the average number of microparticles detected by flow cytometry in all subgroup | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Agnès Charpentier, MD, PhD, Study Director — GHICL
Locations (3):
- France (3):
  - EFS, Lille
  - GHICL, Lille
  - CHRU Lille, Lille

IPD SHARING:
Plan to Share IPD: No